CLINICAL TRIAL: NCT02468635
Title: Analysis of Pulmonary Rehabilitation on the Physical Capacity and Pulmonary Function in Patients With Chronic Obstructive Pulmonary Disease Clinical Trial
Brief Title: Rehabilitation of Patients With Lung Chronic Obstructive Pulmonary Disease
Acronym: PR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Cássio Magalhães da Silva e Silva, Principal Investigator, Federal University of Bahia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ca141078
Record Dates: First submitted 2015-05-30; First posted 2015-06-11 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary rehabilitation; chronic obstructive pulmonary disease; physical ability; pulmonary function; quality of daily life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- without training for upper limb (Other): Receive treatment from traditional pulmonary rehabilitation and without resistive training for upper limb (UL)
  Interventions: Other: without training for upper limb
- upper limb exercises (Other): Receive the same treatment control with additional upper limb resistance training.
  Interventions: Other: upper limb exercises

INTERVENTIONS:
Other: upper limb exercises — HEATING PHASE: diagonals for upper and lower limbs (5-10 minutes). AEROBIC PHASE: aerobic exercise on a treadmill or bicycle between 5 - 30 minutes and rest 1-2 minutes according to the Borg scale and patient tolerance (Borg scores for dyspnea 4-5); RESISTANCE STAGE: upper limb exercises with weight training equipment or dumbbells (the patient's adaptation) with 50% of maximum load reached the maximum repetition test. Series 2 minutes and rest interval between sets 1-2 minutes. RESPIRATORY TRAINING : Strengthening of the respiratory muscles 5-15 minutes with Threshold with load of 50% of the affected MIP (measure maximal inspiratory pressure) evaluation. RELAXATION: Stretching and muscle massage therapy group involved in the 5-10 minute workout.
  Arms: upper limb exercises
Other: without training for upper limb — HEATING PHASE: diagonals for upper and lower limbs (5-10 minutes). AEROBIC PHASE: aerobic exercise on a treadmill or bicycle between 5 - 30 minutes and rest 1-2 minutes according to the Borg scale and patient tolerance (Borg scores for dyspnea 4-5); RESPIRATORY TRAINING: Strengthening respiratory muscles 5-15 minutes with Threshold with load of 50% of MIP hit in the evaluation. RELAXATION: Stretching and muscle massage therapy group involved in the 5-10 minute workout.
  Arms: without training for upper limb

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is characterized by the obstruction is not fully reversible airway, where the severity of the disease and the prognosis is not determined solely by changes in lung function. Pulmonary rehabilitation is a multidisciplinary program of care for patients with chronic respiratory diseases, individually designed to optimize physical and social performance and autonomy of these patients, promoting improvement in functional exercise capacity, quality of life, reducing dyspnea, frequency and duration of hospitalizations and reduce the frequency of exacerbations of the disease. The overall objective of the research is to evaluate the effects of pulmonary rehabilitation program on exercise capacity, lung function, quality of daily life and reduction of dyspnea in patients with COPD. A study type randomized, open-label trial following the recommendations of the CONSORT (Consolidated Standards of Reporting Trials) will be held. The study will be conducted at the Clinic Physiotherapy Course of the School with a sample of 58 patients. The intervention will be performed sessions three times a week for 16 weeks (8 weeks for assessment and 8 weeks for adaptation and (pulmonary rehabilitation training). The PR (pulmonary rehabilitation) will last 60-120 minutes each.O group A (control) will receive treatment of traditional pulmonary rehabilitation and without resistive training for upper limb (UL) and group B will receive the same treatment control with additional training of upper limb strength.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is characterized by the obstruction is not fully reversible airway, where the severity of the disease and the prognosis is not determined solely by changes in lung function. Pulmonary rehabilitation is a multidisciplinary program of care for patients with chronic respiratory diseases, individually designed to optimize physical and social performance and autonomy of these patients, promoting improvement in functional exercise capacity, quality of life, reducing dyspnea, frequency and duration of hospitalizations and reduce the frequency of exacerbations of the disease. It is still reported in the survey improved ability to perform activities of daily life, exercise capacity, quality of life, reduction in respiratory symptoms, anxiety and depression in patients with chronic lung diseases. The overall objective of the research is to evaluate the effects of pulmonary rehabilitation program on exercise capacity, lung function, quality of daily life and reduction of dyspnea in patients with COPD. A study type randomized, open-label trial following the recommendations of the CONSORT (Consolidated Standards of Reporting Trials) will be held. The study will be conducted at the Clinical Department of Physical Therapy School The calculation of the sample held at LEE program (epidemiology laboratory and statistics) with 95% confidence interval and allowing a loss of 20% the sample then goes to 58 patients. Inclusion criteria: Patients with COPD eligible to moderate COPD according to the criteria of gold GOLD (Global Initiative for Chronic Obstructive Lung Disease) as well as being ex-smokers and no exacerbation of the disease in the last three months. Accompanied by a pulmonologist. Age between 40-85 years. Be not practicing physical activity and without cardiovascular or orthopedic disease, make use of bronchodilators and oral theophylline, oxygen therapy or corticosteroids. Exclusion criteria: Patients who have comorbidities musculoskeletal, peripheral saturation of oxygen fall lower than 90% during the 6 minute walk test (six) minutes. Difficulty cognitive understanding of body awareness. The evaluation procedure will be: functional independence measure (FIM); london chest activity of daily living (LCADL); scale medical research council (MRC); the world health organization disability assessment schedule 2.0 (WHODAS 2.0); anthropometric examination; walk test of six (6) minutes; step test; As the repetition maximum (RM); muscle activation - electromyography; grip strength of the upper limbs (DMS); ultrasound diaphragm dynamometer; spirometry; respiratory muscle strength; saint george in respiratory disease questionnaire (SGRQ). The intervention will be performed sessions three times a week for 16 weeks (8 weeks for assessment and 8 weeks for adaptation and PR training). PR will last from 60 to 120 minutes each. Patients who agree to participate and the PR will be divided into two groups randomly through enveloped draw. Group A (control) will receive treatment from traditional pulmonary rehabilitation and without resistive training for upper limb (UL) and group B will receive the same treatment control with additional upper limb resistance training. For data analysis continuous variables will be analyzed with central tendency and dispersion measures, data or dichotomous categorical variables will be analyzed frequently measures. For the realization of inferential statistics are. Since the data are normally distributed, the Student t test for independent samples. The Mann-Whitney test is used to compare the differences in the means of the variables between the groups. To analyze the correlation between the functional capacity variables and QOL will be used in calculating the Pearson correlation coefficient (r) if the data are normally distributed and the calculation of the Spearman correlation coefficient was not distributed normally. To evaluate the reliability will be used the coefficient of intra-class correlation coefficient (ICC). Statistical analysis will be performed using the Statistical Package for Social Sciences for Windows (version 17.0).

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD eligible to moderate COPD according to the criteria of gold GOLD (Global Initiative for Chronic Obstructive Lung Disease) and who had post-bronchodilator spirometry results in the last year of FEV1 (forced expiratory volume in one second) / FVC (forced vital capacity) <0.7 and FEV1 between 50% and 80% of previsto.
* Besides being former smokers for at least three months and were clinically stable, no disease exacerbation in the past three months.
* Accompanied by a pulmonologist.
* Age between 40-85 years.
* They are not practicing physical activity.
* Without cardiovascular or orthopedic disease that makes it impossible to perform the exercises of the RP protocol.
* Without presenting other comorbidities that put them at risk during the exercises .
* Use of bronchodilators and oral theophylline, oxygen therapy or corticosteroids.

Exclusion Criteria:

* Patients who have musculoskeletal comorbidities that interfere with walking or performing upper extremity exercises.
* lower peripheral saturation decrease of oxygen lower than 90% during the 6 minute walk test (six) minutes.
* Presenting difficulty of cognitive understanding of body awareness and the ability to recall information for the questionnaire responses applied in the evaluation and re-evaluation in addition to this also children, adolescents and legally incapable

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-06 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Change in distance of the six-minute walk test | 8 weeks
  measure: metres

SECONDARY OUTCOMES:
Change in quality of life | 8 weeks
  measured by questionnaire Saint George/ measure: points
Change in forced expiratory volume in one second | 8 weeks
  measurement: liters
Change in forced vital capacity | 8 weeks
  measurement: liters
Change in respiratory muscle strength | 8 weeks
  measurement: Water centimeter
repetition maximum (RM); | 8 weeks
  measurement: Kg

CONTACTS AND LOCATIONS:
Overall Officials: Adelmir Machado, research, Study Director — Federal University of Bahia
Locations (1):
- Federal University of Bahia, Salvador, Estado de Bahia, Brazil